CLINICAL TRIAL: NCT03299218
Title: Effectiveness of a Programme Comprised of SNF, Cash-based Transfers and BCC to Prevent Stunting Among Children 6-24 Months in Rahim Yar Khan, Punjab, Pakistan
Brief Title: Effectiveness of SNF, Cash and BCC to Prevent Stunting Among Children 6-24 Months in Rahim Yar Khan, Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Benazir Income Support Programme (BISP) (Other); Punjab Health Care Commission (Other); World Food Programme (WFP) (Unknown)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CBT Study Rahim Yar Khan
Record Dates: First submitted 2017-08-12; First posted 2017-10-03 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Stunting
Keywords: Specialized Nutritious Food (SNF); Social and Behaviour change communication (SBCC); Cash-based transfers
MeSH Terms: conditions — Growth Disorders | interventions — CASP8 and FADD-Like Apoptosis Regulating Protein

STUDY DESIGN:
Intervention Model Description: 1. Control Group
  2. Cash-based transfers only by BISP
  3. Cash-based transfers and Social & behaviour change communication (SBCC)
  4. Cash-based transfer and SNF
  5. Cash-based transfers, SNF and SBCC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Receiving current Government of Punjab health services
- Cash-based transfers (Experimental): Cash-based transfers only by BISP
  Interventions: Other: Cash
- Cash with SBCC (Experimental): Cash-based transfers and Social & behaviour change communication (SBCC)
  Interventions: Behavioral: Social and behaviour change communication (SBCC); Other: Cash
- Cash with SNF (Wawamum) (Experimental): Cash-based transfers and SNF (Wawamum)
  Interventions: Dietary Supplement: SNF (Wawamum); Other: Cash
- Cash,SNF (Wawamum) & SBCC (Experimental): Cash-based transfers, SNF (Wawamum) and SBCC
  Interventions: Dietary Supplement: SNF (Wawamum); Behavioral: Social and behaviour change communication (SBCC); Other: Cash

INTERVENTIONS:
Dietary Supplement: SNF (Wawamum) — A monthly ration of 30 sachets of SNF (one 50 gram sachet of Wawamum per child per day) will be provided by LHWs. Each recruited child will receive SNF on a monthly basis for the duration of 18 months during his/her age of 6-24 months.
  Arms: Cash with SNF (Wawamum); Cash,SNF (Wawamum) & SBCC
Behavioral: Social and behaviour change communication (SBCC) — SBCC messages will be delivered by LHWs in their monthly routine household visits. Male and female group sessions will be arranged on quarterly basis with the help of health committees.
  Arms: Cash with SBCC; Cash,SNF (Wawamum) & SBCC
Other: Cash — Cash totaling 1600 rupees per month will be transferred by BISP throughout the study period.
  Arms: Cash with SBCC; Cash with SNF (Wawamum); Cash,SNF (Wawamum) & SBCC; Cash-based transfers

SUMMARY:
Malnutrition is a public health problem, with long-lasting physiological consequences and increased risk of morbidity and mortality. It can be recognized as one of the key obstacles in national development, due to its influence on individual productivity, school performance and physical work capacity. Malnutrition is a hidden crisis in Pakistan, with rates increasing during the last decade. High prevalence of food insecurity, illiteracy, lack of nutritional knowledge, poor hygiene status, and under recognized role of nutrition are some of the possible causes. The situation of malnutrition in Pakistan necessitates an urgent need for addressing its causes through various nutrition interventions, in order to ensure a bright future for the coming generations.

Although, malnutrition is a major problem across Pakistan, its burden and implications in the remote districts of Punjab are quite evident. The levels of undernutrition in district Rahim Yar Khan are high, with 47% of children being underweight. These numbers also highlight the presence of long-term undernutrition in the district, as evidenced by 45% of the children being stunted in 2014.

Given the alarming situation of child malnutrition in district Rahim Yar Khan, the World Food Program (WFP) Pakistan is proposing an intervention program comprised of cash-based transfers, specialized nutritious foods and behaviours change communication to prevent stunting in district Rahim Yar Khan, province Punjab. The interventions will be delivered through the existing health system and Benazir Income Support Programme (BISP). It is anticipated that the intervention will reduce the widespread macro and micro nutrient malnutrition and food insecurity in the targeted areas. Furthermore, to ensure the presence of adequate evidence to persuade policymakers for further scaling up, it is essential that an impact evaluation be conducted. Therefore, the Department of Paediatrics and Child Health, Aga Khan University (AKU) using robust methodologies on a representative sample size in the district of Rahim Yar Khan to assess the effectiveness of the WFP interventions on process and outcome indicators.

DETAILED DESCRIPTION:
Malnutrition is a public health problem, with long-lasting physiological consequences and increased risk of morbidity and mortality. It can be recognized as one of the key obstacles in national development, due to its influence on individual productivity, school performance and physical work capacity. Malnutrition is a hidden crisis in Pakistan, with rates increasing during the last decade. High prevalence of food insecurity, illiteracy, lack of nutritional knowledge, poor hygiene status, and under recognized role of nutrition are some of the possible causes. The situation of malnutrition in Pakistan necessitates an urgent need for addressing its causes through various nutrition interventions, in order to ensure a bright future for the coming generations.

The second Lancet Series on Maternal and Child Under-nutrition (2013) and the Scaling-Up Nutrition (SUN) Initiative give some recommendations on selected effective approaches for the management and prevention of under-nutrition, such as breastfeeding counselling or micronutrient supplementation, but evidence gaps still remain, particularly concerning indirect interventions. The World Health Organization highlighted in 2010 the need to consider prevention strategies when implementing programs aiming at reducing stunting rates. There is also evidence showing that preventive programs, such as supplementation, can be more effective to reduce childhood under-nutrition than nutrition rehabilitation. Reviews on cash transfer experiences show that this type of intervention has the potential to prevent undernutrition. However, most of the cash transfer programs implemented and scientifically evaluated do not have a clear nutritional objective, which leads to inconclusive evidence regarding their nutritional benefits.

Although, malnutrition is a major problem across Pakistan, its burden and implications in the remote districts of Punjab are especially evident. The levels of undernutrition in district Rahim Yar Khan are high, with 47% of children being underweight. These numbers also highlight the presence of long-term undernutrition in the district, as evidenced by 45% of the children being stunted in 2014.

Given the alarming situation of child malnutrition in Rahim Yar Khan district, the World Food Programme (WFP) Pakistan is proposing an intervention programme comprised of cash-based transfers, specialized nutritious foods and behavior change communication to prevent stunting in Rahim Yar Khan district, Punjab province. The interventions will be delivered through the existing health system and the social protection programme, Benazir Income Support Programme (BISP). It is anticipated that the intervention will reduce the widespread macro and micro nutrient malnutrition and food insecurity in the targeted areas. Furthermore, to ensure the presence of adequate evidence to persuade policymakers for further scaling up, it is essential that an impact evaluation be conducted. The study will be conducted by the Aga Khan University (AKU) using robust methodologies on a representative sample size in the district of Rahim Yar Khan. This document will describe the methods and strategies that AKU will employ to assess the effectiveness of the interventions on process and outcome indicators.

ELIGIBILITY:
Inclusion Criteria:

1. BISP beneficiary for intervention arms and poverty score between 16.18 - 20.00 according to the BISP approach for control group;
2. Living in the catchment area of LHW;
3. Have at least one child of 6-7 months old at the time of inclusion, and;
4. Willing and able to provide written informed consent for the study.

Exclusion Criteria:

1. Non BISP households
2. Planning to migrate form the study area in next 18 months
3. Unable to provide written informed consent
4. Children with severe malnutrition and/or chronic illness

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2179 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Reduction in stunting | 18 months
  10% reduction in stunting in children
SBCC package on the basis of formative research | 3 months
  SBCC package will be developed on the basis of formative research
Cost-effectiveness of intervention packages for prevention of stunting in children | 18 months
  Cost effectiveness analysis will run through the full three years of the program cost

SECONDARY OUTCOMES:
Weight gain in kilograms | 18 months
  Child weight in kilograms will be measured on monthly basis
Length gain in centimeters | 18 months
  Child length in centimeters will be measured on monthly basis
Impact of the intervention on micronutrient deficiencies | At 24 months of age
  Impact of the intervention on micronutrient deficiencies will be measured at 24 months by biochemical analysis
Improvement in IYCF practices | 18 months
  Improvement in IYCF practices will be measured from monthly follow-up data
Improved nutrition, hygiene and health related knowledge and practices | 18 months
  Improved nutrition, hygiene and health related knowledge and practices will be measured from endline KAP data
Proportion of households with moderate or severe hunger (food insecurity) | 18 months
  Food insecurity will be measured from baseline and endline data
Uptake of health services and interventions | 18 months
  Uptake of health services and interventions will be measured from baseline and endline data

CONTACTS AND LOCATIONS:
Overall Officials: Sajid B Soofi, FCPS, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Tehsil Rahim Yar Khan, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Onah MN, Khan GN, Kureishy S, Bourdaire J, de Pee S, Garzon C, Ihtesham Y, Akbar N, Soofi SB. The cost-effectiveness of a cash-based transfer, specialised nutritious food, and social and behaviour change communication intervention package to prevent undernutrition among children 6-23 months in Pakistan: A cluster randomised controlled trial. J Glob Health. 2024 Nov 22;14:04186. doi: 10.7189/jogh.14.04186. PMID 39575728
- [Derived] Soofi SB, Ariff S, Khan GN, Habib A, Kureishy S, Ihtesham Y, Hussain M, Rizvi A, Sajid M, Akbar N, Garzon C, de Pee S, Bhutta ZA. Effectiveness of unconditional cash transfers combined with lipid-based nutrient supplement and/or behavior change communication to prevent stunting among children in Pakistan: a cluster randomized controlled trial. Am J Clin Nutr. 2022 Feb 9;115(2):492-502. doi: 10.1093/ajcn/nqab341. PMID 34612491
- [Derived] Khan GN, Kureishy S, Ariff S, Habib MA, Usmani AA, Mubarik A, Hussain M, Akbar N, Rodriguez de Castro P, Garzon AC, de Pee S, Soofi SB. Specialized Nutritious Food Combined With Cash Transfers and Social and Behavior Change Communication to Prevent Stunting Among Children Aged 6 to 23 Months in Pakistan: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2020 Aug 24;9(8):e19001. doi: 10.2196/19001. PMID 32831183